CLINICAL TRIAL: NCT02888535
Title: Intensive Care Unit and Secondary and Primary Immune Deficiency
Acronym: ICUSPID
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A01246-41
Record Dates: First submitted 2016-05-27; First posted 2016-09-05 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2017-07

CONDITIONS: Primary Immune Deficiency Disorder
Keywords: primary immunodeficiency; secondary immunodeficiency; intensive care unit; infection; adult
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Internal Medicine consultation

SUMMARY:
Primary immune deficiencies (PID) are characterized by a failure of the immune system that is not explained by any infectious, neoplastic, or iatrogenic cause. In 2015, more than 300 different inherited rare disorders were described. The occurrence of PID in adult is rare and diagnosis may be supported by the 6 ESID signs for adult. However these warnings signs are based only on expert recommendations and do not include comprehensive symptoms of PIDs. Recurrent infections, more aggressive, are the most common mode of revelation of the PID. Less frequently, autoimmune manifestation, solid tumor, lymphoproliferation tumor, chronic granulomatosis or hemophagocytic lymphohistiocytosis syndrome (HLS) may also revealed a PID. The objective of this study was to evaluate the occurrence of unknown PID in adult admitted in critical care unit and to determinate if the investigation of PID in patients with severe infections or HLS should be routinely performed in MCIU.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Hospitalized in medical intensive care unit for :
* Severe infection without pathogen identification
* Severe infection due to encapsuled pathogen
* Opportunistic infections or unusual pathogen
* Idiopathic hemophagocytic syndrome

Exclusion Criteria:

* primary immunodeficiency already known
* secondary immunodeficiency already known (HIV, cancer, immunosuppressive or immunomodulatory treatment, nephrotic syndrome, protein-losing enteropathy, severe malnutrition before admission, cirrhosis with hepatic failure, sickle cell disease, splenectomy and moderate chronic renal failure (clearance between 30 and 59 m² min/1.73 ml)
* local-regional factors which can be responsible for infections (history of ear, nose and throat surgery or neurosurgery, history of fracture of the skull base, cystic fibrosis, chronic respiratory insufficient)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 65, hospitalized in medical intensive care unit for a severe or opportunistic infection or an idiopathic hemophagocytic syndrome, without any known warning sign or predisposing factor, were included.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Primary objective : Number of patients with primary immune deficiency diagnosed after an admission in intensive care unit. | A consultation in the Internal Medicine Department is scheduled 3 months after admission in intensive care unit
  A consultation in the Internal Medicine department is schduled 3 months after the hospitalization in intensive care unit to investigate an immune deficiency. This consultation consit on a physical examination and a immune testing. Immune testing included but is not limited to :
  Complete blood count, blood smear Immunoglobulin (Ig) isotype and IgG sub class quantitation (gram per litre) Quantitative serum complement (C3 (milligram per litre), C4 (milligram per litre), CH50 (%) and AP50 when Neisseria meningitides infection) Extensive immunophenotyping of T, B, and natural killer cells (cells/mm3) Specific antibody response to a variety of vaccine (milligram/litre) HIV serology Body computed tomography (CT) scan Lymphocytes, macrophage functional assays or genetic assay when necessary The outcome measure is the number of participants with abnormal laboratory or radiology values leading to primary immune deficiency diagnosis

SECONDARY OUTCOMES:
Secondary objectives : Number of patients diagnosed for a secondary immunodeficiency after admission in intensive care unit | A consultation in the Internal medicine department is scheduled 3 months after admisson in intensive care unit
  A consultation in the Internal Medicine department is schduled 3 months after the hospitalization in intensive care unit to investigate an immune deficiency. This consultation consit on a physical examination and a immune testing. Immune testing included but is not limited to :
  Complete blood count, blood smear Immunoglobulin (Ig) isotype and IgG sub class quantitation (gram per litre) Quantitative serum complement (C3 (milligram per litre), C4 (milligram per litre), CH50 (%) and AP50 when Neisseria meningitides infection) Extensive immunophenotyping of T, B, and natural killer cells (cells/mm3) Specific antibody response to a variety of vaccine (milligram/litre) HIV serology Body computed tomography (CT) scan Lymphocytes, macrophage functional assays or genetic assay when necessary The outcome measure is the number of participants with abnormal laboratory or radiology values leading to secondary immune deficiency diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Martin Silva, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No